CLINICAL TRIAL: NCT04311502
Title: A Phase IIc Trial of Clofazimine- and Rifapentine-Containing Treatment Shortening Regimens in Drug-Susceptible Tuberculosis: The CLO-FAST Study
Brief Title: Clofazimine- and Rifapentine-Containing Treatment Shortening Regimens in Drug-Susceptible Tuberculosis: The CLO-FAST Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual was permanently closed due to futility in the experimental arm on June 22, 2023. Follow-up in the experimental arm was extended to 117 weeks.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5362; 30148 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2020-03-05; First posted 2020-03-17 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: HIV; Tuberculosis
Keywords: rifapentine; clofazimine; drug-susceptible tuberculosis; tuberculosis treatment shortening
MeSH Terms: conditions — Tuberculosis | interventions — rifapentine; Rifampin; Isoniazid; Pyrazinamide; Ethambutol; Clofazimine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Experimental (Experimental): Participants received rifapentine/isoniazid/pyrazinamide/ethambutol (PHZE) + clofazimine (CFZ) 300 mg once daily for 2 weeks; then PHZE + CFZ 100 mg once daily for 6 weeks; then rifapentine/isoniazid/pyrazinamide (PHZ) + CFZ 100 mg once daily for 5 weeks.
  Interventions: Drug: Rifapentine; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol; Drug: Clofazimine loading dose
- Arm 2: Standard of care (Active Comparator): Participants received rifampicin/isoniazid/pyrazinamide/ethambutol (RHZE) for 8 weeks; then rifampicin/isoniazid (RH) for 18 weeks.
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol
- Arm C: PK only subgroup (Experimental): Participants received PHZE + CFZ 100 mg once daily for 4 weeks; then remained on study, and were treated with off study medications according to local SOC (RHZE for 4 weeks; then RH for 18 weeks).
  Interventions: Drug: Rifapentine; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol; Drug: Clofazimine 100 MG

INTERVENTIONS:
Drug: Rifapentine — 1200 mg once daily
  Arms: Arm 1: Experimental; Arm C: PK only subgroup
Drug: Rifampicin — 600 mg once daily
  Arms: Arm 2: Standard of care
Drug: Isoniazid — 300 mg once daily
Drug: Pyrazinamide — 1000mg once daily if weight is 40 to <55kg; 1500mg once daily if weight is 55 to <71kg; 2000mg once if weight is ≥71kg
Drug: Ethambutol — 800 mg once daily if weight is 40 to <55kg; 1200 mg once daily if weight is 55 to <71kg; 1600mg once if weight is ≥71kg
Drug: Clofazimine loading dose — 300 mg once daily for 2 weeks (loading dose), then 100 mg once daily
  Arms: Arm 1: Experimental
Drug: Clofazimine 100 MG — 100 mg once daily
  Arms: Arm C: PK only subgroup

SUMMARY:
The purpose of this study was to compare a 3-month rifapentine (RPT)/clofazimine (CFZ)-containing regimen with a CFZ loading dose with the 6-month standard of care (SOC) regimen for drug-susceptible (DS) tuberculosis (TB).

DETAILED DESCRIPTION:
This study compared a 3-month rifapentine (RPT)/clofazimine (CFZ)-containing regimen with a CFZ loading dose with the 6-month standard of care (SOC) for drug-susceptible (DS) tuberculosis (TB).

Randomization was stratified based on HIV status and the presence of advanced disease as determined by chest X-ray.

Participants were randomized to one of three arms:

* Arm 1 (Experimental): rifapentine/isoniazid/pyrazinamide/ethambutol (PHZE) + CFZ 300 mg once daily for 2 weeks; then PHZE + CFZ 100 mg once daily for 6 weeks; then rifapentine/isoniazid/pyrazinamide (PHZ) + CFZ 100 mg once daily for 5 weeks
* Arm 2 (SOC): rifampicin/isoniazid/pyrazinamide/ethambutol (RHZE) for 8 weeks; then rifampicin/isoniazid (RH) for 18 weeks
* Arm C (PK-only subgroup): PHZE + CFZ 100 mg once daily for 4 weeks; then remain on study, off study medications and treated according to SOC (RHZE for 4 weeks; then RH for 18 weeks)

All participants received pyridoxine (vitamin B6) with each dose of isoniazid (INH) based on current local, national or international dosing guidelines.

Arm 1 participants were treated for 13 weeks (including a 2-week CFZ loading dose of 300 mg daily). Arm 2 participants were treated for 26 weeks, and Arm C participants were treated for 4 weeks.

All participants in Arms 1, 2, and C were followed from randomization to Week 65.

On June 1, 2023, the Data and Safety Monitoring Board (DSMB) recommended that the study permanently close to accrual because of the high rate of treatment failure and TB recurrence. The A5362 team, NIAID and DAIDS leadership, and ACTG leadership concurred with the DSMB's recommendation and the study was closed to accrual on June 2, 2023. A letter of amendment was created that extended follow-up to 117 weeks for some participants in Arm 1.

Due to the early close to accrual, a primary analysis report forming the basis of the primary trial manuscript used data collected at study visits up to and including the date when the last enrolled participant completed the week 26 study visit (September 25. 2023). Another final analysis was performed using data collected at study visits up to the date when the last enrolled participant completed the week 65 assessment.

Study visits included physical examinations; blood, urine, and/or sputum collection; chest X-rays; and electrocardiograms (ECG).

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary TB (among participants with or without history of prior TB treatment) identified within 5 days prior to entry by:

  * At least one sputum specimen positive for M. tuberculosis by molecular TB assay (Xpert) or line probe assay [LPA]) OR
  * At least one sputum specimen positive (1+ or greater) for acid-fast bacilli (AFB) on smear microscopy
  * Note: TB diagnosis for purposes of meeting inclusion criterion can be from a study testing laboratory or from an outside laboratory, as long as it is from a sputum sample collected within 5 days prior to entry.
* Pulmonary TB diagnosed without known INH resistance (e.g., by LPA or Xpert) and without known RIF resistance (e.g., by either LPA or Xpert).
* Absence of HIV-1 infection, as documented by any licensed rapid HIV test or HIV-1 enzyme or chemiluminescence immunoassay (E/CIA) test kit, within 30 days prior to entry OR HIV-1 infection, documented by any licensed rapid HIV test or HIV-1 E/CIA test kit at any time prior to entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen or plasma HIV-1 RNA viral load. Two or more HIV-1 RNA viral loads of >1,000 copies/mL are also acceptable as documentation of HIV-1 infection.
* For participants living with HIV, CD4+ cell count ≥100 cells/mm^3, obtained within 30 days prior to study entry at any network-approved non-US laboratory that is Immunology Quality Assessment (IQA) certified.
* For participants living with HIV must be currently receiving or planning to initiate antiretroviral therapy (ART) at or before study week 8.
* A verifiable address or residence readily accessible to facilitate directly observed therapy (DOT), and willingness to inform the study team of any change of address during the treatment and follow-up period.
* The following laboratory values obtained at or within 5 days prior to entry by any US laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent, or at any network-approved non-US laboratory that operates in accordance with Good Clinical Laboratory Practice (GCLP) and participates in appropriate external quality assurance programs.

  * Serum or plasma alanine aminotransferase (ALT) ≤3 times the upper limit of normal (ULN)
  * Serum or plasma total bilirubin ≤2.5 times ULN
  * Serum or plasma creatinine ≤2 times ULN
  * Serum or plasma potassium ≥3.5 mEq/L and ≤5.5 mEq/L
  * Absolute neutrophil count (ANC) ≥650/mm^3
  * Hemoglobin ≥7.0 g/dL
  * Platelet count ≥50,000/mm^3
* For females of reproductive potential, negative serum or urine pregnancy test within 5 days prior to entry by any US clinic or laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent, or is using a point of care (POC)/CLIA-waived test, or at any network-approved non-US laboratory or clinic that operates in accordance with Good Clinical Laboratory Practice (GCLP) and participates in appropriate external quality assurance programs.
* Female participants of reproductive potential must agree not to participate in the conception process (i.e., active attempt to become pregnant, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, must agree to use at least one reliable nonhormonal method of contraception, as listed below, while on study treatment and for 30 days after stopping study medications.

  * Acceptable forms of contraception include:
  * Condoms
  * Intrauterine device or intrauterine system
  * Cervical cap with spermicide
  * Diaphragm with spermicide
  * Note: Hormonal birth control alone is not acceptable, as it may not be sufficiently reliable in combination with RPT or RIF.
* Female participants who are not of reproductive potential must have documentation of menopause (i.e., at least 1 year amenorrheic), hysterectomy, or bilateral oophorectomy or bilateral tubal ligation.
* Documentation of Karnofsky performance score ≥50 within 30 days prior to entry.
* Documentation of either the presence or absence of advanced disease as determined by chest X-ray within 5 days prior to entry.
* Ability and willingness of participant to provide informed consent.

Exclusion Criteria:

* More than 5 days of treatment directed against active TB for the current TB episode preceding study entry.
* Pregnant or breast-feeding.
* Unable to take oral medications.
* Current receipt of clofazimine or bedaquiline or known receipt of clofazamine or bedaquiline at any time in the past.
* Corrected QT based on the Fridericia correction method (QTcF) interval >450 ms for men or >470 ms for women within 30 days prior to entry.
* Weight <30 kg.
* Current or planned use within 6 months following enrollment of one or more of the following medications: HIV protease inhibitors, HIV entry and fusion inhibitors, HIV non-nucleoside reverse transcriptase inhibitors (other than EFV), elvitegravir/cobicistat, bictegravir, quinidine, procainamide, amiodarone, sotalol, disopyramide, ziprasidone, or terfenadine.
* Current extrapulmonary TB, in the opinion of the site investigator.
* Current or history of known personal or family long QT syndrome.
* Known allergy/sensitivity or any hypersensitivity to components of study TB drugs or their formulation.
* Active drug, alcohol use or dependence; or mental illness (e.g., major depression) that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Known history of acute intermittent porphyria.
* Other medical conditions (e.g., severe uncontrolled diabetes, liver or kidney disease, blood disorders, peripheral neuritis, chronic diarrhea) in which the current clinical condition of the participant is likely to prejudice the response to, or assessment of, treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2025-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Metcalfe, MD, PhD, MPH, Study Chair — University of California, San Francisco
Locations (6):
- Les Centres GHESKIO Clinical Research Site (GHESKIO-INLR) CRS, Port-au-Prince, Haiti
- Byramjee Jeejeebhoy Medical College (BJMC) CRS, Pune, India
- Malawi (2):
  - Malawi CRS, Lilongwe, Central Region
  - Blantyre CRS, Blantyre
- CAPRISA eThekwini CRS, Durban, KwaZulu-Natal, South Africa
- Milton Park CRS, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (ACTG) Network by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the ACTG.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the ACTG Group.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the ACTG "Data Request" form at: https://submit.mis.s-3.net/ Researchers of approved proposals will need to sign an ACTG Data Use Agreement before receiving the data.

REFERENCES:
- [Derived] Mugodhi F, Kanyama C, Makiya F, Metcalfe J, Potani C, Scarsi KK, Weir I, Furin J. "Six months is a lot of time to lie": Anticipated stigma, disclosure and treatment preferences among participants in a tuberculosis therapeutic trial. Res Sq [Preprint]. 2025 Dec 22:rs.3.rs-8277920. doi: 10.21203/rs.3.rs-8277920/v1. PMID 41510291
- [Derived] Metcalfe JZ, Weir IR, Scarsi KK, Mendoza-Ticona A, Pierre S, Hall L, Leon-Cruz J, Svensson EM, Koele SE, Samaneka W, Kanyama C, Yohane M, Nevrekar N, Ntsalaze B, Marc JB, Goth M, Maartens G, Chaisson R; ACTG A5362 study team. A 3-month clofazimine-rifapentine-containing regimen for drug-susceptible tuberculosis versus standard of care (Clo-Fast): a randomised, open-label, phase 2c clinical trial. Lancet Infect Dis. 2026 Jan;26(1):46-54. doi: 10.1016/S1473-3099(25)00436-0. Epub 2025 Sep 4. PMID 40915311
- See also: DAIDS AE Grading Table — https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS — https://rsc.niaid.nih.gov/sites/default/files/manual-exped-aes-v2_0.pdf
- See also: A simple, valid, numerical score for grading chest x-ray severity in adult smear-positive pulmonary tuberculosis — https://thorax.bmj.com/content/65/10/863.long

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from November 2021 to March 2023 in 6 sites located in Malawi (2 sites), South Africa, Zimbabwe, India, and Haiti. A screening and accrual pause was instated on April 4, 2023 and subsequently formally closed to accrual on June 2, 2023 in response to recommendations from the DSMB.
Groups:
- Arm 1: Experimental: Participants received rifapentine/isoniazid/pyrazinamide/ethambutol (PHZE) + clofazimine (CFZ) 300 mg once daily for 2 weeks; then PHZE + CFZ 100 mg once daily for 6 weeks; then rifapentine/isoniazid/pyrazinamide (PHZ) + CFZ 100 mg once daily for 5 weeks.
  Rifapentine: (P) 1200 mg once daily Isoniazid: (H) 300 mg once daily Pyrazinamide: (Z) 1000mg once daily if weight is 40 to <55kg; 1500mg once daily if weight is 55to <71kg; 2000mg once if weight is ≥71kg Ethambutol: (E) 800 mg once daily if weight is 40 to <55kg; 1200 mg once daily if weight is 55 to <71kg; 1600mg once if weight is ≥71kg Clofazimine loading dose: (CFZ) 300 mg once daily for 2 weeks (loading dose), then 100 mg once daily
- Arm 2: Standard of Care: Participants received rifampicin/isoniazid/pyrazinamide/ethambutol (RHZE) for 8 weeks; then rifampicin/isoniazid (RH) for 18 weeks.
  Rifampicin: (R) 600 mg once daily Isoniazid: (H) 300 mg once daily Pyrazinamide: (Z) 1000mg once daily if weight is 40 to <55kg; 1500mg once daily if weight is 55to <71kg; 2000mg once if weight is ≥71kg Ethambutol: (E) 800 mg once daily if weight is 40 to <55kg; 1200 mg once daily if weight is 55 to <71kg; 1600mg once if weight is ≥71kg
- Arm C: PK Only Subgroup: Participants received PHZE + CFZ 100 mg once daily for 4 weeks; then remained on study, and were treated with off study medications according to local SOC (RHZE for 4 weeks; then RH for 18 weeks).
  Rifapentine: (P) 1200 mg once daily Isoniazid: (H) 300 mg once daily Pyrazinamide: (Z) 1000mg once daily if weight is 40 to <55kg; 1500mg once daily if weight is 55to <71kg; 2000mg once if weight is ≥71kg Ethambutol: (E) 800 mg once daily if weight is 40 to <55kg; 1200 mg once daily if weight is 55 to <71kg; 1600mg once if weight is ≥71kg Clofazimine: (CFZ) 100 mg once daily
Period: Overall Study
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care | Arm C: PK Only Subgroup
Started | 58 | 31 | 15
Started Treatment and Were Not Late Exclusions | 55 | 31 | 15
Completed | 22 | 27 | 14
Not Completed | 36 | 4 | 1
Not completed — Death | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 3 | 0
Not completed — Participant is in prison | 1 | 0 | 0
Not completed — Participant moved out of country | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — DSMB Mandated Extension of follow-up | 29 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care | Arm C: PK Only Subgroup | Total
Number analyzed (Participants) | 58 | 31 | 15 | 104
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [27 to 39] | 30 [24 to 38] | 35 [31 to 43] | 33 [27 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 2 | 22
  Male | 47 | 22 | 13 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 49 | 26 | 15 | 90
  Unknown or Not Reported | 9 | 5 | 0 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN | 9 | 6 | 0 | 15
  BLACK OR AFRICAN AMERICAN | 49 | 25 | 15 | 89
Region of Enrollment [Number; unit: participants]
  Haiti | 2 | 2 | 0 | 4
  India | 9 | 5 | 0 | 14
  Malawi | 26 | 11 | 9 | 46
  South Africa | 11 | 6 | 3 | 20
  Zimbabwe | 10 | 7 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Time to 12 Weeks Stable Culture Conversion in Liquid Media
Description: The time of stable culture conversion was the visit corresponding to the first of two consecutive negative cultures without an intervening positive, and/or visits wherein the participant was unable to produce sputum and had no signs of active TB.
  If a participant did not culture convert, they were censored at their last culture result (regardless of result). If a participant died before conversion they were censored at 12 weeks. Participants who were lost to follow-up prior to 12 weeks with their last culture being positive were censored at 12 weeks (i.e. assumed they did not have a culture conversion by week 12), and participants who were lost to follow-up prior to 12 weeks with their last culture being negative were censored at the last sampling visit for which they had a valid culture result.
Time Frame: From Entry through Week 12
Population: Efficacy set: All participants who were randomized to study treatment Arm 1 or Arm 2 and were not late exclusions.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 55 | 31
weeks | 6 [4 to 8] | 8 [6 to 10]
Statistical Analysis 1: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; This comparison is adjusting for HIV-1 status (positive/negative) and TB Disease at Screening (Advanced/Not Advanced); Test type: Superiority; p = 0.21, Regression, Cox; Adjusted for HIV-1 status (positive/negative) and TB Disease at Screening (Advanced/Not Advanced); Hazard Ratio (HR) = 1.21, 90% CI 2-sided [0.82 to 1.79] — Arm 1 vs Arm 2

2. Primary Outcome: Participants Experiencing Any Grade 3 or Higher Adverse Event (AE) That is at Least a One Grade Increase From Baseline Over 65 Weeks
Description: An adverse event is any unfavorable and unintended sign, symptom, or diagnosis that occurs in a study participant during the conduct of the study REGARDLESS of the attribution.
  Adverse events are graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death. AE grading was per Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table V2.1, Corrected Version 2.1, July 2017)
  The primary manuscript outcome measure includes data through week 65 up to September 25, 2023
Time Frame: From entry through Week 65
Population: Safety set: All participants who started assigned study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care | Arm C: PK Only Subgroup
Number analyzed (Participants) | 58 | 31 | 15
Participants
  Number of Participants through Primary Manuscript Cutoff date of September 25, 2023 | 26 | 5 | 3
  Number of Participants through Week 65 | 27 | 6 | 3
Statistical Analysis 1: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; The point estimate and 90% two-sided confidence intervals for the difference in cumulative proportions of participants experiencing a Grade 3 or higher AE that is at least one-grade increase from baseline at any time during the 65-week study period was compared between Arm 1 and Arm 2. This outcome measure is limited to data obtained up to September 25, 2023; Test type: Superiority; p < 0.01, Wald chi-square test; Risk Difference (RD) = 0.30, 90% CI 2-sided [0.14 to 0.45] — Difference in cumulative proportions (Arm 1 - Arm 2)
Statistical Analysis 2: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; The point estimate and 90% two-sided confidence intervals for the difference in cumulative proportions of participants experiencing a Grade 3 or higher AE that is at least one-grade increase from baseline at any time during the 65-week study period was compared between Arm 1 and Arm 2. All data through week 65; Test type: Superiority; p < 0.01, Wald chi-square test; Risk Difference (RD) = 0.28, 90% CI 2-sided [0.11 to 0.44] — Difference in cumulative proportions (Arm 1 - Arm 2)

3. Secondary Outcome: Proportion of Participants With Favorable Clinical/Bacteriologic Outcome (Definition A) at 65 Weeks Post-randomization
Description: Favorable Outcome are:
  * liquid culture negative at week 65
  * without signs or symptoms of ongoing active TB and unable to produce sputum at 65 weeks
  * who at the end of the follow-up period are clinically without signs/symptoms of ongoing active TB and produce a sputum specimen that is contaminated in two liquid cultures without evidence of TB
  Unfavorable:
  * Absence of cure: Having a sputum sample at or after EOT that is culture-positive (any medium) with a second positive sample obtained 4 hours following the first sample.
  * Death from any cause except for violent or accidental cause
  * Had a positive culture for Mtb when last seen
  * Had a treatment extension beyond nominal level due to clinically inadequate response
  Unevaluable are:
  * lost to follow-up during treatment or post-treatment with their last culture being negative for Mtb
  * violent or accidental death
  * becoming pregnant during their assigned active treatment and stop their assigned treatment.
Time Frame: From entry through Week 65
Population: Efficacy set: All participants who were randomized to study treatment Arm 1 or Arm 2 and were not late exclusions.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 55 | 31
proportion of participants | .50 [0.35 to 0.62] | .76 [.56 to .88]
Statistical Analysis 1: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; The point estimate and 95% two-sided confidence interval for the difference in cumulative proportions of participants experiencing a favorable outcome through week 65 was compared between Arm 1 and Arm 2; Test type: Superiority; p = 0.01, Wald chi-square test; Risk Difference (RD) = -0.26, 95% CI 2-sided [-0.47 to -0.06] — Difference in cumulative proportions (Arm 1 - Arm 2)

4. Secondary Outcome: Proportion of Participants With Favorable Composite Outcome (Definition B) at 65 Weeks Post-randomization
Description: Favorable Outcome are:
  Same as definition A
  Unfavorable:
  Same as definition A and:
  * lost to follow-up during treatment phase
  * failing to complete treatment
  * receiving any one or more of the following: extension of treatment beyond the nominal level, except to make up missed doses; re-starting treatment following >= 30 consecutive days lost to follow-up; a change in at least one drug in treatment regimen for any reason except re-infection, pregnancy, or temporary drug challenge
  Unevaluable are:
  * lost to follow-up after treatment phase, and not assessable at the end of follow-up, with their last culture being negative for Mtb
  * Violent death or accidental death
  * Women who become pregnant during their assigned active treatment and stop their assigned treatment
Time Frame: From entry through Week 65
Population: Efficacy set: All participants who were randomized to study treatment Arm 1 or Arm 2 and were not late exclusions.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 55 | 31
proportion of participants | 0.49 [0.35 to 0.61] | 0.74 [0.54 to 0.86]
Statistical Analysis 1: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.02, Wald chi-square; Risk Difference (RD) = -0.25, 95% CI 2-sided [-0.46 to -0.04] — Difference in cumulative proportions (Arm 1 - Arm 2)

5. Secondary Outcome: Number of Participants Who Prematurely Discontinue Their Treatment Regimen Through 65 Weeks
Description: Premature discontinuation is defined as discontinuation other than due to violent death, natural disaster, or administrative censoring
Time Frame: From entry through Week 65
Population: Safety set: All participants who started assigned study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 55 | 31
Participants | 2 | 3
Statistical Analysis 1: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; Test type: Superiority — Fisher's exact test was used to test for a difference in proportions; p = 0.35, Fisher Exact; Risk Difference (RD) = -0.06, 95% CI 2-sided [-0.22 to 0.05] — Difference in proportions (Arm 1 - Arm 2); exact confidence interval

6. Secondary Outcome: Mean QTcF
Description: QT interval measured as the average of three electrocardiogram (ECG) readings taken 5-10 minutes apart, corrected with Fridericia correction
Time Frame: Measured at Weeks 2, 8, and 13 (end of investigational treatment)
Population: Limited to available data
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 58 | 31
ms
  Mean QTcF Interval at Week 2: number analyzed (Participants) | 56 | 29
  Mean QTcF Interval at Week 2 | 419 (19.4) | 401 (14.8)
  Mean QTcF Interval at Week 8: number analyzed (Participants) | 54 | 31
  Mean QTcF Interval at Week 8 | 422 (16.8) | 408 (16.8)
  Mean QTcF Interval at Week 13: number analyzed (Participants) | 55 | 30
  Mean QTcF Interval at Week 13 | 427 (19.5) | 407 (20.4)

7. Secondary Outcome: QTcF Interval Mean Change From Baseline
Description: Mean change from baseline in mean QTcF at weeks 2, 8, and end of treatment (EOT)
Time Frame: Measured at baseline and Weeks 2, 8, and 13 (end of investigational treatment)
Population: Limited to participants with available data
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 58 | 31
ms
  Change in mean QTcF from Week 2 to Screening: number analyzed (Participants) | 56 | 29
  Change in mean QTcF from Week 2 to Screening | 23.9 (21.2) | 0.736 (19.8)
  Change in mean QTcF from Week 8 to Screening: number analyzed (Participants) | 54 | 31
  Change in mean QTcF from Week 8 to Screening | 26.5 (20.1) | 7.38 (14.6)
  Change in mean QTcF from Week 13 to Screening: number analyzed (Participants) | 55 | 30
  Change in mean QTcF from Week 13 to Screening | 31.6 (20.7) | 7.77 (19.0)
Statistical Analysis 1: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; Test type: Superiority; p < 0.01, Regression, Linear; GEE = 24.04, 95% CI 2-sided [15.13 to 32.94]

8. Secondary Outcome: Categorized QTcF
Description: Absolute QTcF was categorized as:< 480; ≥480 ms and <500 ms; ≥500 ms
Time Frame: Week 2, 8, and Week 13
Population: Safety set: participants who started Arm 1 and Arm 2 and with data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 58 | 31
Participants
  Week 2: number analyzed (Participants) | 56 | 29
  Week 2: Absolute QTcF ≥480 ms and <500 ms | 0 | 0
  Week 2: Absolute QTcF ≥500 ms | 0 | 0
  Week 2: Absolute QTcF < 480 ms | 56 | 29
  Week 8: number analyzed (Participants) | 54 | 31
  Week 8: Absolute QTcF ≥480 ms and <500 ms | 0 | 0
  Week 8: Absolute QTcF ≥500 ms | 0 | 0
  Week 8: Absolute QTcF < 480 ms | 54 | 31
  Week 13: number analyzed (Participants) | 55 | 30
  Week 13: Absolute QTcF ≥480 ms and <500 ms | 0 | 0
  Week 13: Absolute QTcF ≥500 ms | 0 | 0
  Week 13: Absolute QTcF < 480 ms | 55 | 30

9. Secondary Outcome: Categorized Change From Baseline
Description: Categorized change from baseline as: change from baseline of <30 ms; change from baseline of ≥30 ms and <60 ms; change from baseline of ≥60 ms
Time Frame: Measured at Weeks 2, 8, and Week 13
Population: Limited to the safety analysis set, participants who started assigned treatment, in Arm 1 and Arm 2 and with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 58 | 31
Participants
  Week 2: number analyzed (Participants) | 56 | 29
  Week 2: QTcF change from baseline of ≥30 ms and <60 ms | 15 | 1
  Week 2: QTcF change from baseline of ≥60 ms | 2 | 0
  Week 2: QTcF change from baseline of <30 ms | 39 | 28
  Week 8: number analyzed (Participants) | 54 | 31
  Week 8: QTcF change from baseline of ≥30 ms and <60 ms | 17 | 2
  Week 8: QTcF change from baseline of ≥60 ms | 1 | 0
  Week 8: QTcF change from baseline of <30 ms | 36 | 29
  Week 13: number analyzed (Participants) | 55 | 30
  Week 13: QTcF change from baseline of ≥30 ms and <60 ms | 22 | 3
  Week 13: QTcF change from baseline of ≥60 ms | 5 | 0
  Week 13: QTcF change from baseline of <30 ms | 28 | 27
Statistical Analysis 1: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; Compares the odds of participants having maximum occurrence of QTcF change from baseline of ≥30 ms and <60 ms, or ≥60 ms between Arm 1 and Arm 2 in the safety set using the proportional odds model; Test type: Superiority; p < 0.01, Regression, Logistic; Odds Ratio (OR) = 7.15, 95% CI 2-sided [2.40 to 21.30]
Statistical Analysis 2: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; Proportion of Participants with Worst Changes in QTcF from Screening >= 30 ms over visits at Weeks 2, 8, 13; Test type: Superiority; p < 0.01, exact unconditional; Risk Difference (RD) = 0.41, 95% CI 2-sided [0.17 to 0.58] — Arm 1 - Arm 2

10. Secondary Outcome: Time to Stable Culture Conversion in Liquid Media Through Week 65
Description: Defined as the first of two (consecutive or non-consecutive) negative sputum cultures without an intervening positive culture, and/or visits wherein the participant is unable to produce sputum and has no signs of active TB
Time Frame: From entry through Week 65
Population: Efficacy set: All participants who were randomized to study treatment Arm 1 or Arm 2 and were not late exclusions.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 55 | 31
weeks | 6 [4 to 8] | 8 [6 to 10]
Statistical Analysis 1: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; Test type: Superiority; p = 0.18, Regression, Cox — One-sided p-value; Adjusted for HIV status (positive/negative) and TB disease according to chest X-ray (advanced/not advanced); Hazard Ratio (HR) = 1.23, 90% CI 2-sided [0.84 to 1.80] — Arm 1 vs. Arm 2

11. Secondary Outcome: Time to Stable Culture Conversion in Solid Media Through Week 65
Description: The time of stable culture conversion was the visit corresponding to the first of two consecutive negative cultures without an intervening positive, and/or visits wherein the participant was unable to produce sputum and had no signs of active TB.
  If a participant did not culture convert, they were censored at their last culture result (regardless of result). If a participant died before conversion, the death was considered as a competing event. Participants who were lost to follow-up prior to 65 weeks with their last culture being positive were censored at 65 weeks (i.e. assumed they did not have a culture conversion by week 65), and participants who were lost to follow-up prior to 65 weeks with their last culture being negative were censored at the last sampling visit for which they had a valid culture result.
  Adjusted model adjusts for HIV-1 status (positive/negative) and TB Disease at Screening (Advanced/Not Advanced).
Time Frame: From entry through Week 65
Population: Efficacy set: All participants who were randomized to study treatment Arm 1 or Arm 2 and were not late exclusions.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 55 | 31
weeks | 6 [2 to 8] | 6 [4 to 8]
Statistical Analysis 1: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; This comparison is adjusting for HIV-1 status (positive/negative) and TB Disease at Screening (Advanced/Not Advanced); Test type: Superiority; p = 0.25, Regression, Cox — One-sided p-value; Hazard Ratio (HR) = 1.17, 90% CI 2-sided [0.80 to 1.71]

12. Secondary Outcome: Number of Participants Achieving Stable Liquid Culture Conversion by Week 8
Description: as for outcome 10
Time Frame: From entry through Week 8
Population: Efficacy set: All participants who were randomized to study treatment Arm 1 or Arm 2 and were not late exclusions.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 55 | 31
Participants | 41 | 19
Statistical Analysis 1: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; Test type: Superiority; p = 0.23, Fisher Exact; Risk Difference (RD) = 0.13, 95% CI 2-sided [-0.07 to 0.35]

13. Secondary Outcome: Number of Participants Achieving Stable Solid Culture Conversion by Week 8
Description: as for outcome 10
Time Frame: From entry through Week 8
Population: Efficacy set: All participants who were randomized to study treatment Arm 1 or Arm 2 and were not late exclusions.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 55 | 31
Participants | 47 | 25
Statistical Analysis 1: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; Test type: Superiority; p = 0.56, Fisher Exact; Risk Difference (RD) = 0.05, 95% CI 2-sided [-0.11 to 0.24]

14. Secondary Outcome: Number of Participants With One or More Serious Adverse Events (SAEs)
Description: Cumulative proportion with at least one Serious Adverse Event (SAE)
  A SAE is defined as any untoward medical occurrence that:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Is an important medical event that many not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the other outcomes listed in the definition above.
Time Frame: From entry through Week 65
Population: Safety set: All participants who started assigned study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care | Arm C: PK Only Subgroup
Number analyzed (Participants) | 58 | 31 | 15
Participants | 8 | 2 | 2
Statistical Analysis 1: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; The point estimate and 90% two-sided confidence intervals for the difference in cumulative proportions of participants experiencing an SAE through week 65 was compared between Arm 1 and Arm 2; Test type: Superiority; p = 0.27, Wald chi-square test; Risk Difference (RD) = 0.07, 90% CI 2-sided [-0.04 to 0.18] — Difference in cumulative proportions (Arm 1 - Arm 2)

15. Secondary Outcome: Number of Participants Achieving Stable Solid Culture Conversion by Week 12
Description: as for outcome 10
Time Frame: From entry through Week 12
Population: Efficacy set: All participants who were randomized to study treatment Arm 1 or Arm 2 and were not late exclusions.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 55 | 31
Participants | 53 | 30
Statistical Analysis 1: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; Test type: Superiority — Fisher's exact test was used to test for a difference in proportions; p = 1, Fisher Exact; Risk Difference (RD) = -0, 95% CI 2-sided [-0.10 to 0.13] — Difference in proportions (Arm 1 - Arm 2); exact confidence interval

16. Secondary Outcome: Median Time (Days) to Positivity in Liquid Culture (MGIT)
Description: Time (days) to positivity in liquid culture (MGIT) is defined as the number of days it takes for the culture to produce results up to a max of 42 days. For negative culture results, time to positivity is imputed as 42 days.
Time Frame: From screening, entry, weeks 1, 2, 3, 4, 6, 8, 10, 12
Population: Efficacy set: All participants who were randomized to study treatment Arm 1 or Arm 2 and were not late exclusions with data available.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 55 | 31
days
  Screening Time to Positivity | 6.17 [3.83 to 7.67] | 5.67 [4.04 to 8.08]
  Entry Time to Positivity: number analyzed (Participants) | 55 | 30
  Entry Time to Positivity | 8.63 [6.67 to 11.2] | 8.23 [7.21 to 10.3]
  Week 1 Time to Positivity: number analyzed (Participants) | 19 | 0
  Week 1 Time to Positivity | 12.8 [7.33 to 18.3] |
  Week 2 Time to Positivity: number analyzed (Participants) | 54 | 29
  Week 2 Time to Positivity | 16.8 [11.8 to 22.4] | 12.1 [9.96 to 18.9]
  Week 3 Time to Positivity: number analyzed (Participants) | 19 | 0
  Week 3 Time to Positivity | 20.2 [8.29 to 42] |
  Week 4 Time to Positivity: number analyzed (Participants) | 54 | 31
  Week 4 Time to Positivity | 25.1 [16.8 to 42] | 16.5 [14.4 to 38]
  Week 6 Time to Positivity: number analyzed (Participants) | 51 | 30
  Week 6 Time to Positivity | 42 [27.2 to 42] | 42 [17.6 to 42]
  Week 8 Time to Positivity: number analyzed (Participants) | 50 | 29
  Week 8 Time to Positivity | 42 [42 to 42] | 42 [26.7 to 42]
  Week 10 Time to Positivity: number analyzed (Participants) | 52 | 29
  Week 10 Time to Positivity | 42 [42 to 42] | 42 [42 to 42]
  Week 12 Time to Positivity: number analyzed (Participants) | 52 | 30
  Week 12 Time to Positivity | 42 [42 to 42] | 42 [42 to 42]
Statistical Analysis 1: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; Time point: Screening; Test type: Superiority; p = 0.597, Regression, Cox; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.57 to 1.39]
Statistical Analysis 2: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; Time point: Entry; Test type: Superiority; p = 0.70, Regression, Cox; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.58 to 1.44]
Statistical Analysis 3: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; Time point: Week 2; Test type: Superiority; p = 0.07, Regression, Cox; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.40 to 1.03]
Statistical Analysis 4: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; Time point: Week 4; Test type: Superiority; p = 0.04, Regression, Cox; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.34 to 0.98]
Statistical Analysis 5: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; Time point: Week 6; Test type: Superiority; p = 0.60, Regression, Cox; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.41 to 1.67]
Statistical Analysis 6: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; Time point: Week 8; Test type: Superiority; p = 0.595, Regression, Cox; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.33 to 1.88]
Statistical Analysis 7: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; Time point: Week 10; Test type: Superiority; p = 0.66, Regression, Cox; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.25 to 2.44]
Statistical Analysis 8: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; Time point: Week 12; Test type: Superiority; p = 0.86, Regression, Cox; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.21 to 6.39]

17. Secondary Outcome: Change in Chest X-ray Score From Baseline to End of Treatment in Each Arm
Description: The chest X-ray was posterior-anterior. Extent of disease (limited to one lobe or region, unilateral, bilateral, or diffuse) and cavitation status (cavities present [location] or absent) was documented by validated numerical score (percent of total lung affected by any pathology + 40 if cavitation is present; 0 = No percent affected, 140 = entire lung is affected + cavitation is present) for grading chest X-ray in adult smear-positive pulmonary TB (Thorax 2010; 65(10):863-9).
  Analysis was conducted based on site readings of CXR
Time Frame: Entry, End of Treatment (Week 13 for Arm 1 and Week 26 for Arm 2)
Population: Efficacy set: All participants who were randomized to study treatment Arm 1 or Arm 2 and were not late exclusions and had data available at both time points.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 53 | 29
score on a scale | -25.51 [-34.27 to -16.75] | -46.10 [-58.04 to -34.16]
Statistical Analysis 1: Comparison: Arm 1: Experimental vs Arm 2: Standard of Care; This comparison is adjusting for HIV-1 status (positive/negative) and TB Disease at Screening (Advanced/Not Advanced); Test type: Superiority; p < 0.01, Regression, Linear; Slope = 20.43, 95% CI 2-sided [5.71 to 35.16]

18. Secondary Outcome: Proportion of Participants Who Have a TB Relapse, From End of Treatment Until Week 65
Description: The time of relapse is defined as the time from end of treatment until the first sputum sample that is culture positive in liquid or solid media for an Mtb strain that has matching genotype with the baseline isolate (as determined by whole genome sequencing). A second positive sputum sample obtained at least 4 hours following the first sputum collection is required to confirm a relapse. If the second sputum sample was negative, this was not counted as a relapse. If a participant was lost to follow-up without a second sputum sample confirmation of relapse (including contaminated or missing), it was counted as a relapse.
  Whole genome sequencing of samples, which is necessary to assess TB relapse, was not performed due to lack of funding. There is no plan to test these samples in the future.
Time Frame: From end of treatment (week 13 for Arm 1; week 26 for Arm 2) to week 65
Population: No participants have results as results for whole genome sequencing, which is necessary to assess TB relapse, was not performed due to lack of funding. There is no plan to test these samples in the future.
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Cumulative Proportion of Participants Who Have a TB Recurrence, From End of Treatment Until Week 65
Description: The time of recurrence is defined as the time from end of treatment until the first sputum sample that is culture positive in liquid or solid media. A second positive sputum sample obtained at least 4 hours following the first sputum collection is required to confirm a recurrence. If the second sputum sample was negative, this will not be counted as a recurrence. If a participant was lost to follow-up without a second sputum sample confirmation of recurrence (including contaminated or missing), it was counted as a recurrence.
  Participants at risk for recurrence where those who were stable culture conversions by end of treatment.
Time Frame: From end of treatment (week 13 for Arm 1; week 26 for Arm 2) to week 65
Population: Efficacy set: All participants who were randomized to study treatment Arm 1 or Arm 2 and were not late exclusions and at risk for TB Recurrence
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 48 | 29
proportion of participants
  Within 26 Weeks of Treatment Completion | 0.21 [0.12 to 0.35] | 0.04 [0.01 to 0.24]
  Within 39 Weeks of Treatment Completion | 0.23 [0.13 to 0.37] | 0.04 [0.01 to 0.24]
  Within 52Weeks of Treatment Completion: number analyzed (Participants) | 48 | 0
  Within 52Weeks of Treatment Completion | 0.23 [0.13 to 0.37] |

20. Secondary Outcome: Pharmacokinetic Parameter for CFZ: Minimum Concentration (Cmin)
Description: Estimated using noncompartmental methods applied to concentrations from intensive PK sampling visits at weeks 2 and 13.
Time Frame: Measured at Weeks 2 and 13
Population: Intensive PK tests were performed at weeks 2 and 13 on Arm 1 participants who consent and were registered to the Intensive PK subgroup and at week 2 on Arm C participants.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Arm 1: Experimental | Arm C: PK Only Subgroup
Number analyzed (Participants) | 19 | 15
mg/L
  Week 2: number analyzed (Participants) | 18 | 15
  Week 2 | 0.473 (0.181) | 0.169 (0.088)
  Week 13: number analyzed (Participants) | 17 | 0
  Week 13 | 0.594 (0.197) |

21. Secondary Outcome: Pharmacokinetic Parameter for CFZ: Maximum Concentration (Cmax)
Description: Estimated using noncompartmental methods applied to concentrations from intensive PK sampling visits at weeks 2 and 13.
Time Frame: Measured at Weeks 2 and 13
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Arm 1: Experimental | Arm C: PK Only Subgroup
Number analyzed (Participants) | 19 | 15
mg/L
  Week 2: number analyzed (Participants) | 18 | 15
  Week 2 | 0.861 (0.286) | 0.277 (0.123)
  Week 13: number analyzed (Participants) | 17 | 0
  Week 13 | 0.819 (0.247) |

22. Secondary Outcome: Pharmacokinetic Parameter for CFZ: Time of Cmax (Tmax)
Description: Estimated using noncompartmental methods applied to concentrations from intensive PK sampling visits at weeks 2 and 13.
Time Frame: Measured at Weeks 2 and 13
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm 1: Experimental | Arm C: PK Only Subgroup
Number analyzed (Participants) | 19 | 15
hours
  Week 2: number analyzed (Participants) | 18 | 15
  Week 2 | 4.97 (2.10) | 7.74 (4.90)
  Week 13: number analyzed (Participants) | 17 | 0
  Week 13 | 7.27 (4.68) |

23. Secondary Outcome: Pharmacokinetic Parameter for CFZ: Area Under the Concentration Curve (AUC0-24h)
Description: Estimated using noncompartmental methods applied to concentrations from intensive PK sampling visits at weeks 2 and 13.
Time Frame: Measured at Weeks 2 and 13
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mg/L*h
Arm/Group | Arm 1: Experimental | Arm C: PK Only Subgroup
Number analyzed (Participants) | 19 | 15
mg/L*h
  Week 2: number analyzed (Participants) | 18 | 15
  Week 2 | 15.6 (5.58) | 5.42 (2.48)
  Week 13: number analyzed (Participants) | 17 | 0
  Week 13 | 16.9 (5.57) |

24. Secondary Outcome: Mean Change From Baseline in Skin Pigmentation (Colorimetric L*)
Description: The median of triplicate measurements of Inner Arm, and Face (median of all measurements from the Chin, Forehead, Left Cheek, and Right Cheek). L represents lightness (0 = black, 100 = white).
  Further data processing removed values if one of the triplicates differed more than 5% of the median.
Time Frame: Entry, Weeks 8, 13, 26, and 65
Population: Limited to the safety analysis set, participants who started assigned treatment, and were not premature study discontinuations before week 8 and had data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 55 | 30
units on a scale
  Inner Arm - Week 8: number analyzed (Participants) | 49 | 24
  Inner Arm - Week 8 | -2.54 (2.51) | -1.65 (2.17)
  Inner Arm - Week 13: number analyzed (Participants) | 47 | 26
  Inner Arm - Week 13 | -4.72 (3.1) | 0.02 (2.74)
  Inner Arm - Week 26: number analyzed (Participants) | 47 | 25
  Inner Arm - Week 26 | -2.8 (3) | -0.68 (2.54)
  Inner Arm - Week 65: number analyzed (Participants) | 46 | 24
  Inner Arm - Week 65 | -1.15 (3.45) | 1.19 (3.52)
  Face - Week 8: number analyzed (Participants) | 54 | 30
  Face - Week 8 | -3 (2.30) | -0.96 (2.16)
  Face - Week 13 | -3.61 (2.86) | -0.51 (1.97)
  Face - Week 26: number analyzed (Participants) | 53 | 29
  Face - Week 26 | -2.65 (2.5) | -0.43 (2.16)
  Face - Week 65: number analyzed (Participants) | 49 | 26
  Face - Week 65 | -0.45 (2.96) | 0.34 (2.31)

25. Secondary Outcome: Mean Change From Baseline in Skin Pigmentation (Colorimetric a*)
Description: The median of triplicate measurements of Inner Arm, and Face (median of all measurements from the Chin, Forehead, Left Cheek, and Right Cheek). The a* parameter represents the balance between red and green. Positive values of a* indicate a reddish tone, while negative values indicate a greenish tone. (-128 = Green, 127 = Red).
  Further data processing removed values if one of the triplicates differed more than 5% of the median.
Time Frame: Entry, Weeks 8, 13, 26, and 65
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 55 | 30
units on a scale
  Inner Arm - Week 8: number analyzed (Participants) | 49 | 24
  Inner Arm - Week 8 | 0.23 (5.86) | .20 (2.44)
  Inner Arm - Week 13: number analyzed (Participants) | 47 | 26
  Inner Arm - Week 13 | 2.14 (8.61) | -0.34 (6.40)
  Inner Arm - Week 26: number analyzed (Participants) | 47 | 25
  Inner Arm - Week 26 | -1.09 (5.72) | -1.01 (4.97)
  Inner Arm - Week 65: number analyzed (Participants) | 46 | 24
  Inner Arm - Week 65 | -0.96 (5.51) | -1.37 (5.96)
  Face - Week 8: number analyzed (Participants) | 53 | 30
  Face - Week 8 | -0.58 (1.86) | -0.09 (3.77)
  Face - Week 13: number analyzed (Participants) | 54 | 30
  Face - Week 13 | -0.46 (2.99) | -0.28 (1.19)
  Face - Week 26: number analyzed (Participants) | 52 | 29
  Face - Week 26 | -0.66 (1.71) | -0.43 (1.56)
  Face - Week 65: number analyzed (Participants) | 49 | 26
  Face - Week 65 | -0.23 (2.20) | 0.23 (2.01)

26. Secondary Outcome: Mean Change From Baseline in Skin Pigmentation (Colorimetric b*)
Description: The median of triplicate measurements of Inner Arm, and Face (median of all measurements from the Chin, Forehead, Left Cheek, and Right Cheek). The b* parameter represents the balance between yellow and blue. Positive values of b* indicate a yellowish tone, while negative values indicate a bluish tone (-128 = Blue, 127 = Yellow).
  Further data processing removed values if one of the triplicates differed more than 5% of the median.
Time Frame: Entry, Weeks 8, 13, 26, and 65
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 55 | 30
units on a scale
  Inner Arm - Week 8: number analyzed (Participants) | 49 | 24
  Inner Arm - Week 8 | -1.62 (3.49) | -1.21 (3.07)
  Inner Arm - Week 13: number analyzed (Participants) | 47 | 26
  Inner Arm - Week 13 | -2.27 (3.38) | 0.11 (4.28)
  Inner Arm - Week 26: number analyzed (Participants) | 47 | 25
  Inner Arm - Week 26 | -1.52 (4.50) | -0.71 (3.86)
  Inner Arm - Week 65: number analyzed (Participants) | 46 | 24
  Inner Arm - Week 65 | -1.70 (3.37) | -1.29 (4.06)
  Face - Week 8: number analyzed (Participants) | 54 | 30
  Face - Week 8 | -2.48 (2.15) | -0.82 (2.97)
  Face - Week 13 | -2.65 (2.75) | -0.66 (2.44)
  Face - Week 26: number analyzed (Participants) | 53 | 29
  Face - Week 26 | -2.44 (2.89) | -0.92 (2.55)
  Face - Week 65: number analyzed (Participants) | 49 | 26
  Face - Week 65 | -1.72 (2.52) | -0.88 (2.17)

27. Secondary Outcome: Change From Baseline in Participant-reported Changes in Skin Pigment Related to Perceived Skin Hyperpigmentation
Description: Subjective questionnaire asked the following questions :
  1.) On a scale from 0 to 10: (0 being none and 10 being most significant possible) How would you rate any change in the coloration of your skin since you began TB treatment?
Time Frame: Entry, Weeks 8, 13, 26, and 65
Population: Participants in Arm 1 and Arm 2 with follow-up after week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 55 | 30
score on a scale
  Week 8 | 1.60 (2.65) | 0.53 (1.11)
  Week 13: number analyzed (Participants) | 55 | 29
  Week 13 | 2.15 (2.65) | 0.17 (0.54)
  Week 26: number analyzed (Participants) | 53 | 29
  Week 26 | 0.53 (1.41) | 0.79 (1.95)
  Week 65: number analyzed (Participants) | 52 | 26
  Week 65 | 0.25 (1.60) | 0.38 (1.68)

28. Secondary Outcome: Change From Baseline in Participant-reported Distress Caused by Change in Skin Pigment Related to Perceived Skin Hyperpigmentation
Description: Subjective questionnaire asked the following questions:
  On a scale from 0 to 10: (0 being none and 10 being worst possible) How would you rate your distress to skin coloration changes since you began TB treatment, if any?
Time Frame: Entry, Weeks 8, 13, 26, and 65
Population: Participants in Arm 1 and Arm 2 with follow-up after week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Experimental | Arm 2: Standard of Care
Number analyzed (Participants) | 55 | 30
score on a scale
  Week 8 | 1.02 (2.48) | 0.17 (0.75)
  Week 13: number analyzed (Participants) | 55 | 29
  Week 13 | 0.89 (2.01) | -0.07 (0.26)
  Week 26: number analyzed (Participants) | 53 | 29
  Week 26 | 0.21 (1.52) | 0.07 (0.80)
  Week 65: number analyzed (Participants) | 52 | 26
  Week 65 | 0.21 (1.70) | 0.15 (0.88)

ADVERSE EVENTS:
Time Frame: From entry through Week 65
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, July 2017. An adverse event is any unfavorable and unintended sign, symptom, or diagnosis that occurs in a study participant during the conduct of the study REGARDLESS of the attribution.
  Adverse events are graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death.
Groups:
- Arm1: Participants received rifapentine/isoniazid/pyrazinamide/ethambutol (PHZE) + clofazimine (CFZ) 300 mg once daily for 2 weeks; then PHZE + CFZ 100 mg once daily for 6 weeks; then rifapentine/isoniazid/pyrazinamide (PHZ) + CFZ 100 mg once daily for 5 weeks.
  Doses (administered orally once daily): rifapentine, 1200mg; isoniazid, 300mg; pyrazinamide, 40 to <55kg 1000mg, 55to <71kg 1500mg; ≥71kg 2000mg; ethambutol, 40 to <55kg 800mg, 55to <71kg 1200mg; ≥71 kg 1600mg
  Rifapentine: 1200 mg once daily
  Isoniazid: 300 mg once daily
  Pyrazinamide: 1000mg once daily if weight is 40 to <55kg 1500mg once daily if weight is 55to <71kg 2000mg once if weight is ≥71kg
  Ethambutol: 800 mg once daily if weight is 40 to <55kg 1200 mg once daily if weight is 55 to <71kg 1600mg once if weight is ≥71kg
  Clofazimine: 300 mg once daily for 2 weeks (loading dose). 100 mg once daily
- Arm2: Participants received rifampicin/isoniazid/pyrazinamide/ethambutol (RHZE) for 8 weeks; then rifampicin/isoniazid (RH) for 18 weeks.
  Doses (administered orally once daily): rifampicin, 600mg; isoniazid, 300mg; pyrazinamide, 40 to <55kg 1000mg, 55to <71kg 1500mg; ≥71 kg 2000mg; ethambutol, 40 to <55kg 800mg, 55to <71kg 1200mg; ≥71 kg 1600mg
  Rifampicin: 600 mg once daily
  Isoniazid: 300 mg once daily
  Pyrazinamide: 1000mg once daily if weight is 40 to <55kg 1500mg once daily if weight is 55to <71kg 2000mg once if weight is ≥71kg
  Ethambutol: 800 mg once daily if weight is 40 to <55kg 1200 mg once daily if weight is 55 to <71kg 1600mg once if weight is ≥71kg
- ArmC: Participants received PHZE + CFZ 100 mg once daily for 4 weeks; then remained on study, and were treated with off study medications according to local SOC (RHZE for 4 weeks; then RH for 18 weeks).
  Doses (for on study medications; administered orally once daily): rifapentine, 1200mg; isoniazid, 300mg; pyrazinamide, 40 to <55kg 1000mg, 55to <71kg 1500mg; ≥71 kg 2000mg; ethambutol, 40 to <55kg 800mg, 55to <71kg 1200mg; ≥71 kg 1600mg
  Rifapentine: 1200 mg once daily
  Isoniazid: 300 mg once daily
  Pyrazinamide: 1000mg once daily if weight is 40 to <55kg 1500mg once daily if weight is 55to <71kg 2000mg once if weight is ≥71kg
  Ethambutol: 800 mg once daily if weight is 40 to <55kg 1200 mg once daily if weight is 55 to <71kg 1600mg once if weight is ≥71kg
  Clofazimine: 300 mg once daily for 2 weeks (loading dose). 100 mg once daily
Arm/Group | Arm1 | Arm2 | ArmC
All-Cause Mortality (participants affected / at risk) | 1/58 | 1/31 | 1/15
Serious Adverse Events (participants affected / at risk) | 8/58 | 2/31 | 2/15
Other Adverse Events (participants affected / at risk) | 25/58 | 7/31 | 3/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm1 (N=58) | Arm2 (N=31) | ArmC (N=15)
Cor pulmonale (Cardiac disorders) | 1 | 0 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Ocular icterus (Hepatobiliary disorders) | 1 | 0 | 0
Cerebral toxoplasmosis (Infections and infestations) | 0 | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 1
Immune reconstitution inflammatory syndrome associated tuberculosis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm1 (N=58) | Arm2 (N=31) | ArmC (N=15)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0
Scabies (Infections and infestations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1
Blood albumin decreased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 14 | 3 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Glycosuria (Renal and urinary disorders) | 1 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Enrollment to this study was terminated early based on a recommendation from the independent DSMB for the study. This was due to the high rate of unfavorable outcomes and recurrences in Arm 1. As a consequence, the study had reduced precision to evaluate the primary biomarker outcome related to time to stable culture conversion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (4):
  • Study Protocol and Informed Consent Form: Protocol Version 2.0 (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT04311502/Prot_ICF_000.pdf
  • Study Protocol: Clarification Memo 1 (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT04311502/Prot_001.pdf
  • Study Protocol: Letter of Amendment 1 (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT04311502/Prot_002.pdf
  • Statistical Analysis Plan (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT04311502/SAP_003.pdf